CLINICAL TRIAL: NCT01191645
Title: Can Opioid Induced Effects on Esophageal Motility and Lower Esophageal Sphincter be Counteracted by a Dopamine Receptor Antagonist?
Brief Title: Opioid Effects on Swallowing and Esophageal Sphincter Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Johanna Savilampi, MD, Region Örebro County
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: JS002
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Opioid Induced Pharyngeal and Esophageal Dysfunction
Keywords: Lower esophageal sphincter pressure; Esophageal motility; Remifentanil; Metoclopramide; Naloxone; High resolution solid state manometry
MeSH Terms: conditions — Esophageal Diseases | interventions — Naloxone; Remifentanil; Sodium Chloride; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Primperan (Experimental)
  Interventions: Drug: metoclopramide
- Naloxon (Active Comparator)
  Interventions: Drug: naloxone
- Natriumklorid (Placebo Comparator)
  Interventions: Drug: Sodium Chloride
- Ultiva (Experimental)
  Interventions: Drug: remifentanil

INTERVENTIONS:
Drug: naloxone — Injection fluid, solution 0,4 mg/kg Bolus infusion 6ug/kg at one occasion Continuous infusion 0,1 ug/kg/minute during 50 min
  Other Names: Naloxon; ACT-code: V03AB15
  Arms: Naloxon
Drug: remifentanil — Powder for injection/ infusion fluid solution, 2 mg Infusion TCI 1ng/kg 10 min ( 0,05 ug/kg/min) Infusion TCI 2ng/kg 10 min ( 0.10 ug/kg/min) Infusion TCI 3ng/kg 20 min ( 0,15 ug/kg/min)
  Other Names: Ultiva; ATC-code: N01AH06
  Arms: Ultiva
Drug: Sodium Chloride — Infusion fluid, solution 9 mg/ml ( hydrogenic solution )
  Other Names: Natriumklorid; ACT-code: B05XA03
  Arms: Natriumklorid
Drug: metoclopramide — Injection fluid, solution 5 mg/mg Iv injection 0,2 mg/kg at one occasion
  Other Names: Primperan
  Arms: Primperan

SUMMARY:
The purpose of this study is to determine whether a dopamine receptor antagonist metoclopramide can counteract opioid induced effects on esophageal motility and lower esophageal sphincter. The aim of this study is also to evaluate if the opioid antagonist naloxone reduces the opioid induced pharyngeal and esophageal dysfunction.

DETAILED DESCRIPTION:
Opioids induce pharyngeal and esophageal dysfunction and reduce the lower esophageal sphincter (LES) pressure, and thereby decreases the barrier pressure between the stomach and esophagus. This contributes to an increased risk of regurgitation and aspiration during anaesthesia induction and in the postoperative period, when the patient is treated with opioids for pain relief.

The effect of opioid antagonists on the opioid induced pharyngeal dysfunction and lower esophageal sphincter pressure are unknown. In a recently performed clinical trial we found that the peripheral opioid antagonist methylnaltrexone didn't have effect on the pharyngeal induced pharyngeal and esophageal dysfunction.This indicates that the negative opioid induced effects are not peripherally induced or mediated via peripheral opioid receptors.

In previously performed studies most of the volunteers reported swallowing problems when receiving infusion of the opioid remifentanil, we have also found that remifentanil abolished spontaneous esophageal motility.

The purpose of the study is to evaluate if opioid induced effects on the lower esophageal sphincter can be counteracted by a dopamine receptor antagonist, metoclopramide. It is previously known that dopamine, a catecholamine neurotransmitter, decreases the lower esophageal sphincter pressure and that a dopamine antagonist has the ability to increase the pressure.

Further in this study we want to evaluate if the opioid antagonist naloxone, which affects both peripheral and central opioid receptors, reduces the opioid induced pharyngeal and esophageal dysfunction.

A third aim of the study is to evaluate if the previously reported swallowing difficulties during infusion of opioid remifentanil are dose related, consequently does a higher concentration of opioids increase the swallowing difficulties.

The pharyngeal and esophageal motility/function can be registered in an easy and objective way with the high resolution manometry, ManoScan 360. ManoScan 360 is an equipment with 36 sensors at 1 cm spacing with 12 tip transducers at every sensor. The 36 closely spaced sensors automatically capture all relevant motor function from the pharynx to the stomach. The system collects reliable and consistent data records with improved diagnostic accuracy, and the data are analyzed using ManoView analyzes software. ManoScan 360 has a CE mark approval and has been used at Örebro University Hospital during the last three years.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 40 year old healthy volunteers from both sexes.
2. Have signed and dated Informed Consent.
3. Willing and able to comply with the protocol for the duration of the trial.

Exclusion Criteria:

1. Anamnesis of pharyngoesophageal dysfunction
2. Known history of cardiac, pulmonary or neurological disease
3. Ongoing medication
4. Allergies to or history of reaction to naloxone, remifentanil, fentanyl analogues or metoclopramide
5. Pregnancy or breast feeding
6. BMI > 30
7. Previous participation in a medical clinical trial where opioid has been used or have during last 30 days participated in any other medicinal clinical trial or in a trial where follow-up in not completed.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Lower esophageal sphincter pressure | 2 hours

SECONDARY OUTCOMES:
Swallowing difficulties | 2 hours
  The volunteers will be asked to do dry swallowing and assess the swallowing difficulty on the basis of following criteria: no difficulties, mild, moderate or severe difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Wattwil, MD, Principal Investigator — University Hospital Örebro
Locations (1):
- Örebro University Hospital, Örebro, Sweden